CLINICAL TRIAL: NCT04180657
Title: Investigation of Ghrelin Levels in Patients With Protein C Deficiency
Brief Title: Ghrelin Levels in Patients With Protein C Deficiency
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 69965
Record Dates: First submitted 2019-10-21; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-10

CONDITIONS: Protein C Deficiency
Keywords: ghrelin; growth hormone; protein C deficiency; appetite
MeSH Terms: conditions — Protein C Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with protein C deficiency: Patient and control group are compared regarding ghrelin, growth hormone levels and appetite, and no other intervention is made.
  Interventions: Genetic: Protein C deficiency
- Healthy controls: Patient and control group are compared regarding ghrelin, growth hormone levels and appetite, and no other intervention is made.

INTERVENTIONS:
Genetic: Protein C deficiency — The effect of protein C deficiency on ghrelin levels are investigated.
  Groups: Patients with protein C deficiency

SUMMARY:
In rodents with protein C deficiency elevated levels of ghrelin has been observed. The purpose of this study is to investigate if patients with protein C deficiency also have elevated levels of ghrelin, and if so, how this affects the patients.

30 patients with protein C deficiency and 30 healthy BMI and gender matched controls are recruited. Bloodsamples are taken in order to measure ghrelin and GH levels and other metabolic parameters. The patients and controls are also asked to answer a questionaire regarding appetite.

If patients with protein C deficiency have higher levels of ghrelin than the general population, this will lead to new studies that will perhaps help us understand the importance of ghrelin in humans.

ELIGIBILITY:
Inclusion Criteria:

* protein C deficiency or healthy subjects
* age 18-70
* BMI 18-35
* written statement to join the study

Exclusion Criteria:

* chronic illness, apart from protein C deficiency and lifestyle diseases
* everyday medication apart from statins, oral diabetes medication and antihypertensive drugs.
* blood donation within three months prior to the investigation.
* Alcohol abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with protein C deficiency and gender and BMI matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
acyl ghrelin and des acyl ghrelin measured in mg/dl | 6 month

SECONDARY OUTCOMES:
Growth hormone measured in pmol/L | 6 month

IPD SHARING:
Plan to Share IPD: No